CLINICAL TRIAL: NCT00349167
Title: A Phase I, Multi-Center, Open Label, Dose Escalation Trial of the Safety and Pharmacokinetics of Intravenous PR-104 Given Every 3 Weeks in Patients With Solid Tumors
Brief Title: PR-104 in Treating Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Proacta, Incorporated (Industry)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PR104-1001; P30CA016042 (NIH); UCLA-0512034-01A; PROACTA-PR-104-1001
Record Dates: First submitted 2006-07-05; First posted 2006-07-06 (Estimated); Last update posted 2012-11-30 (Estimated); Status verified 2012-11

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — PR-104

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PR-104 (Experimental): PR104 was administered as a 1-hr IV infusion every 21 days at doses ranging from 135 to 1400 mg/m2
  Interventions: Drug: PR-104; Other: laboratory biomarker analysis; Other: pharmacological study

INTERVENTIONS:
Drug: PR-104
Other: laboratory biomarker analysis
Other: pharmacological study

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as PR-104, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing.

PURPOSE: This phase I trial is studying the side effects and best dose of PR-104 in treating patients with advanced solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Evaluate the safety and tolerability of PR-104 in patients with advanced solid tumors.
* Determine the maximum tolerated dose of PR-104 in these patients.

Secondary

* Characterize the pharmacokinetics of PR-104 and its alcohol metabolite in these patients.
* Assess evidence of antitumor activity of this drug in these patients.

Tertiary

* Examine metabolic changes in tumors of these patients using fludeoxyglucose F 18 positron emission tomography scanning.

OUTLINE: This is a multicenter, open-label, prospective, uncontrolled, dose-escalation study.

Patients receive PR-104 IV over 60 minutes on day 1. Treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of PR-104 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

Blood is collected at baseline and then periodically during study treatment for pharmacokinetic and tumor marker studies. Patients undergo fludeoxyglucose F 18 positron emission tomography scanning before beginning study treatment and after completion of course 2 to assess metabolic activity of the tumor.

After completion of study treatment, patients are followed at 30 days.

PROJECTED ACCRUAL: A total of 30 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed solid tumor, meeting 1 of the following criteria:

  * Not amenable to standard therapy
  * Refractory to conventional therapy
* Measurable or evaluable disease

PATIENT CHARACTERISTICS:

* Karnofsky performance status 70-100%
* Life expectancy > 3 months
* Absolute neutrophil count ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Hemoglobin > 9 g/L (transfusion independent)
* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* ALT and AST ≤ 2.5 times ULN
* Creatinine clearance ≥ 60 mL/min
* PT/INR or aPTT ≤ 1.1 times ULN
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 30 days after completion of study treatment
* No significant cardiac comorbidity including any of the following:

  * New York Heart Association class III-IV congenital heart failure
  * LVEF < 40%
  * Unstable angina
  * Myocardial infarction within the past 6 months
  * Ventricular arrhythmias requiring drug therapy
  * Pacemaker or implanted defibrillator
* No ongoing coagulopathy
* No uncontrolled infection or infection requiring parenteral antibiotics
* No other significant clinical disorder or laboratory finding that would preclude study treatment
* No known HIV positivity
* No known positivity for hepatitis B surface antigen or hepatitis C with abnormal liver tests
* No known allergy to nonplatinum-containing alkylating agents

PRIOR CONCURRENT THERAPY:

* Recovered from prior therapy
* More than 2 weeks since prior hormonal therapy (except for androgen-deprivation therapy)
* More than 4 weeks since prior major surgery
* More than 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin C)
* More than 4 weeks since prior radiotherapy
* More than 1 month since prior investigational drugs, therapies, or devices
* No prior radiotherapy to > 25% of bone marrow
* No prior high-dose chemotherapy, either myeloablative or nonmyeloablative (mini-allogeneic transplant)
* No more than 3 prior myelosuppressive chemotherapy regimens
* Concurrent steroids allowed provided dose is stable for ≥ 2 weeks and clinical condition is stable for 1 month

  * Nasal, opthalmologic, and topical glucocorticoid preparations allowed
  * Physiologic hormone replacement therapies allowed (i.e., oral replacement glucocorticoid therapy for adrenal insufficiency)
* No concurrent prophylactic hematopoietic growth factors
* No concurrent radiotherapy, including local palliative radiotherapy or systemic radioisotopes

  * Radioisotopes for protocol specified positron emission tomography allowed
* No other concurrent investigational agents
* No other concurrent chemotherapy, radiotherapy (including palliative local radiotherapy), hormonal therapy (except for androgen-deprivation therapy), and/or biological therapy (including immunotherapy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2005-12; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark D. Pegram, MD, Principal Investigator — Jonsson Comprehensive Cancer Center
Locations (1):
- Jonsson Comprehensive Cancer Center at UCLA, Los Angeles, California, United States

REFERENCES:
- [Result] Jameson MB, Rischin D, Pegram M, Gutheil J, Patterson AV, Denny WA, Wilson WR. A phase I trial of PR-104, a nitrogen mustard prodrug activated by both hypoxia and aldo-keto reductase 1C3, in patients with solid tumors. Cancer Chemother Pharmacol. 2010 Mar;65(4):791-801. doi: 10.1007/s00280-009-1188-1. Epub 2009 Dec 10. PMID 20012293